CLINICAL TRIAL: NCT06813651
Title: Safety, Tolerability and Efficacy of Adjunctive TBO-309 in Reperfusion for Stroke With Tandem Occlusion
Acronym: Co-STARS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ThromBio Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Co-STARS; Application No. 00039 (Other Grant/Funding Number: NSW Biosciences Fund 2023 [2023 NSW BioSF])
Record Dates: First submitted 2025-01-21; First posted 2025-02-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Tandem Occlusion
Keywords: Ischaemic stroke; Stenting; Endovascular thrombectomy; tandem occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, open-label, Bayesian Optimal Phase 2 (BOP2) trial.
  Two intervention doses will be tested sequentially for TBO-309, with 60mg tested first. Then either a higher (120mg) or lower (30mg) dose will be tested, based on results of the 60 mg dose.
  The maximum number of subjects is estimated to be 78 in this two-dose BOP2 design study.
Who Masked: Outcomes Assessor
Masking Description: Masking Description:
  Independent imaging assessors will review and adjudicate blinded study data to ensure the primary endpoint meets consistent pre-determined diagnostic criteria.
  Imaging assessors will be qualified physicians who are independent of the study and not involved in study management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TBO-309 - 60 mg (Experimental): An intravenous (IV) bolus of TBO-309 will be administered before the acute stent procedure. The allocated dose of TBO-309 will be given IV as follows:
  20% of the dose will be administered as a bolus over approximately one minute; then the remainder of the dose (80%) will be administered over 3 hours as an infusion.
  Interventions: Drug: TBO-309: 60 mg
- TBO-309 - 120 mg (Experimental): An intravenous (IV) bolus of TBO-309 will be administered before the acute stent procedure. The allocated dose of TBO-309 will be given IV as follows:
  20% of the dose will be administered as a bolus over approximately one minute; then the remainder of the dose (80%) will be administered over 3 hours as an infusion.
  Interventions: Drug: TBO-309: 120 mg
- TBO-309 - 30 mg (Experimental): An intravenous (IV) bolus of TBO-309 will be administered before the acute stent procedure. The allocated dose of TBO-309 will be given IV as follows:
  20% of the dose will be administered as a bolus over approximately one minute; then the remainder of the dose (80%) will be administered over 3 hours as an infusion.
  Interventions: Drug: TBO-309: 30 mg

INTERVENTIONS:
Drug: TBO-309: 60 mg — TBO-309 is a potent, selective and ATP competitive PI3Kβ inhibitor which blocks platelet activation adhesion/aggregation and promotes platelet disaggregation. By targeting PI3Kβ, TBO-309 specifically inhibits thrombosis whilst minimizing the impact on normal haemostasis.
  Arms: TBO-309 - 60 mg
Drug: TBO-309: 120 mg — TBO-309 is a potent, selective and ATP competitive PI3Kβ inhibitor which blocks platelet activation adhesion/aggregation and promotes platelet disaggregation. By targeting PI3Kβ, TBO-309 specifically inhibits thrombosis whilst minimizing the impact on normal haemostasis.
  Arms: TBO-309 - 120 mg
Drug: TBO-309: 30 mg — TBO-309 is a potent, selective and ATP competitive PI3Kβ inhibitor which blocks platelet activation adhesion/aggregation and promotes platelet disaggregation. By targeting PI3Kβ, TBO-309 specifically inhibits thrombosis whilst minimizing the impact on normal haemostasis.
  Arms: TBO-309 - 30 mg

SUMMARY:
Co-STAR is a multicenter, prospective, open-label, Bayesian Optimal Phase 2 (BOP2) trial that aims to assess the safety and efficacy of adjunctive intravenous TBO-309 in Acute Ischaemic Stroke (AIS) patients with tandem occlusion receiving intra-cranial endovascular thrombectomy (EVT) and acute extracranial carotid artery stenting.

Co-STARS study will test the hypothesis that patients with tandem occlusion treated with EVT and acute stenting in conjunction with TBO-309 will:

* have persistent stent patency without requiring rescue therapy with GPIIb/IIIa inhibitors and
* not experience high rates of symptomatic intra-cranial haemorrhage (sICH).

Patients with tandem occlusion undergoing EVT and acute stenting will receive intravenous TBO-309 bolus and infusion. TBO-309 is a potent, selective and ATP competitive PI3K[beta] inhibitor which reduces platelet activation adhesion/aggregation particularly under conditions of disturbed blood flow and promotes platelet disaggregation. By targeting PI3K[beta], TBO-309 specifically inhibits thrombosis whilst minimizing the impact on normal hemostasis.

DETAILED DESCRIPTION:
Stroke due to large vessel occlusion (LVO) typically causes large infarcts and results in severe disability and a high case fatality rate. Treating LVO by thrombectomy poses technical challenges, especially when the lesion involves not only the extracranial (cervical) part of the internal carotid artery but also its concomitant intracranial distal segment or the ipsilateral middle cerebral artery (tandem occlusion). For patients with tandem occlusion, stenting of the internal carotid is considered acceptable, but it requires the use of antiplatelet therapy to avoid stent thrombosis, often necessitating rescue therapy with GPIIb/IIIa inhibitors. This can lead to an increased risk of hemorrhage especially when potent antiplatelet agents such as GPIIb/IIIa inhibitors are used.

The novel investigational agent TBO-309 is a potent, selective and ATP competitive PI3K[beta] inhibitor which reduces platelet activation adhesion/aggregation particularly under conditions of disturbed blood flow and promotes platelet disaggregation. By targeting PI3K[beta], TBO-309 specifically inhibits thrombosis whilst minimizing the impact on normal hemostasis. This study aims to assess the safety and efficacy of adjunctive TBO-309 in acute ischaemic stroke with tandem occlusion eligible to undergo intra-cranial EVT and acute extracranial carotid artery stenting.

The primary endpoint of this trial is a composite outcome of efficacy and safety, defined by:

1. Avoidance of intra-procedural GPIIb/IIIa inhibitor rescue therapy due to stent thrombosis, combined with persistent stent patency seen on angiographic imaging at 24-36 hours, and
2. no sICH.

This trial will use Bayesian Optimal Phase 2 (BOP2) trial design, and two intervention doses will be tested sequentially for TBO-309. TBO-309 at the dose of 60 mg will be tested first. Then either a higher dose of 120 mg or a lower dose of 30 mg will be tested based on the results of the 60 mg dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or more
2. Patient has an AIS due to tandem occlusion, including large vessel occlusion (LVO) within the intra-cranial anterior circulation and presumed atherosclerotic occlusion of the cervical internal carotid artery origin
3. CT perfusion indicates the presence of salvageable brain tissue, defined as ischaemic core <70mL with a mismatch ratio >1.8 and absolute mismatch >15mL.
4. Patient has at least a mild grade of neurological impairment (NIHSS >4)
5. Patient has an estimated pre-stroke mRS of less than 4

Exclusion Criteria:

1. Patient is considered unlikely to benefit from study intervention defined by one of the following:

   1. Advanced dementia
   2. Severe pre-stroke disability (mRS score 4-5)
   3. Glasgow Coma Score (GCS) 3 to 5
   4. Evidence of a large well-defined ischaemic lesion measuring more than one third of the middle cerebral artery (MCA) territory
2. Uncontrolled hypertension (SBP >180 or DBP >110, refractory to medical therapy)
3. Intracranial haemorrhage within the last 90 days
4. Myocardial infarction or stroke within the last 30 days
5. Patient has an underlying disease process with a life expectancy of <90 days
6. Known treatment with anticoagulants
7. Known severe liver disease
8. Known bleeding disorder
9. Cardiopulmonary resuscitation or arterial puncture at non-compressible site or lumbar puncture within 7 days
10. Another medical illness or social circumstance that may interfere with outcome assessments and follow-up
11. Known or suspected pregnancy
12. Patients currently participating in another interventional clinical trial
13. Informed consent unable to be obtained from the patient or their Person Responsible/Medical Treatment Decision Maker prior to study interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a composite outcome of efficacy and safety | 24-36 hours
  The primary endpoint is a composite outcome of efficacy and safety, defined by the proportion of patients who 1) avoid intra-procedural GPIIb/IIIa inhibitor rescue therapy due to stent thrombosis, combined with persistent stent patency seen on angiographic imaging at 24-36 hours, and 2) have no sICH. sICH is defined as parenchymal haemorrhage type 2 (PH2) on imaging.

SECONDARY OUTCOMES:
Proportion of patients achieving reperfusion. | 24 hours
  The proportion of patients achieving reperfusion, where reperfusion is defined by the expanded Thrombolysis in Cerebral Infarction scale (eTICI) 2b50 or better (i.e. 50% to 100%)
Infarct volume 24-36 hours post study drug commencement | 24-36 hours
Proportion of all patients with any ICH within 24-36 hours post study drug commencement | 24-36 hours
  All ICH as demonstrated on brain imaging at 24-36 hours, where ICH will be classified according to The Heidelberg Bleeding Classification.
Proportion of patients experiencing any bleeding within 24-36 hours of study drug commencement. | 24-36 hours
  The proportion of patients experiencing any bleeding within 24-36 hours of study drug commencement. Bleeding will be determined using a modified WHO scale with grades 1 and 2 classified as minor bleeding, and grades 3 and 4 as major bleeding.
National Institutes of Health Stroke Scale (NIHSS) at 24 hours, and 7 days/at hospital Discharge | 24 hours and 7 days
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurological examination stroke scale. Scores range from 0 to 42, with higher scores indicating greater severity.
Modified Rankin Scale (mRS) score at discharge and 90 days | 90 days
  The Modified Rankin Scale (mRS) is a scale from 0 to 6, with higher scores indicating greater disability (5), and death (6).
Proportion of patients with all-cause mortality at 90 days. | 90 days

OTHER OUTCOMES:
Proportion of patients with sICH | 24-36 hours
  The safety outcome is symptomatic intra-cranial haemorrhage (sICH) within 24-36 hours of study drug commencement. sICH is defined as parenchymal haemorrhage type 2 (PH2) on imaging within 24-36 hours after treatment, associated with a ≥ four-point deterioration on the National Institutes of Health Stroke Scale (NIHSS) from baseline or from the lowest score to 24-36 hours or leading to death.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Miteff - Interventional Neurologist, RACP, CCINR, Principal Investigator — John Hunter Hospital, Newcastle, NSW Australia
Locations (2):
- Australia (2):
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saver JL, Chaisinanunkul N, Campbell BCV, Grotta JC, Hill MD, Khatri P, Landen J, Lansberg MG, Venkatasubramanian C, Albers GW; XIth Stroke Treatment Academic Industry Roundtable. Standardized Nomenclature for Modified Rankin Scale Global Disability Outcomes: Consensus Recommendations From Stroke Therapy Academic Industry Roundtable XI. Stroke. 2021 Aug;52(9):3054-3062. doi: 10.1161/STROKEAHA.121.034480. Epub 2021 Jul 29. PMID 34320814
- [Background] Miller AB, Hoogstraten B, Staquet M, Winkler A. Reporting results of cancer treatment. Cancer. 1981 Jan 1;47(1):207-14. doi: 10.1002/1097-0142(19810101)47:13.0.co;2-6. PMID 7459811
- [Background] Heddle NM, Cook RJ, Tinmouth A, Kouroukis CT, Hervig T, Klapper E, Brandwein JM, Szczepiorkowski ZM, AuBuchon JP, Barty RL, Lee KA; SToP Study Investigators of the BEST Collaborative. A randomized controlled trial comparing standard- and low-dose strategies for transfusion of platelets (SToP) to patients with thrombocytopenia. Blood. 2009 Feb 12;113(7):1564-73. doi: 10.1182/blood-2008-09-178236. Epub 2008 Dec 24. PMID 19109560
- [Background] von Kummer R, Broderick JP, Campbell BC, Demchuk A, Goyal M, Hill MD, Treurniet KM, Majoie CB, Marquering HA, Mazya MV, San Roman L, Saver JL, Strbian D, Whiteley W, Hacke W. The Heidelberg Bleeding Classification: Classification of Bleeding Events After Ischemic Stroke and Reperfusion Therapy. Stroke. 2015 Oct;46(10):2981-6. doi: 10.1161/STROKEAHA.115.010049. Epub 2015 Sep 1. No abstract available. PMID 26330447
- [Background] Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kuelkens S, Larrue V, Lees KR, Roine RO, Soinne L, Toni D, Vanhooren G; SITS-MOST investigators. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet. 2007 Jan 27;369(9558):275-82. doi: 10.1016/S0140-6736(07)60149-4. PMID 17258667
- [Background] Jackson SP, Schoenwaelder SM. Antithrombotic phosphoinositide 3-kinase beta inhibitors in humans: a 'shear' delight! J Thromb Haemost. 2012 Oct;10(10):2123-6. doi: 10.1111/j.1538-7836.2012.04912.x. No abstract available. PMID 22943292
- [Background] Nylander S, Wagberg F, Andersson M, Skarby T, Gustafsson D. Exploration of efficacy and bleeding with combined phosphoinositide 3-kinase beta inhibition and aspirin in man. J Thromb Haemost. 2015 Aug;13(8):1494-502. doi: 10.1111/jth.13027. Epub 2015 Jul 23. PMID 26096765
- [Background] Nylander S, Kull B, Bjorkman JA, Ulvinge JC, Oakes N, Emanuelsson BM, Andersson M, Skarby T, Inghardt T, Fjellstrom O, Gustafsson D. Human target validation of phosphoinositide 3-kinase (PI3K)beta: effects on platelets and insulin sensitivity, using AZD6482 a novel PI3Kbeta inhibitor. J Thromb Haemost. 2012 Oct;10(10):2127-36. doi: 10.1111/j.1538-7836.2012.04898.x. PMID 22906130
- [Background] Jackson SP, Schoenwaelder SM, Goncalves I, Nesbitt WS, Yap CL, Wright CE, Kenche V, Anderson KE, Dopheide SM, Yuan Y, Sturgeon SA, Prabaharan H, Thompson PE, Smith GD, Shepherd PR, Daniele N, Kulkarni S, Abbott B, Saylik D, Jones C, Lu L, Giuliano S, Hughan SC, Angus JA, Robertson AD, Salem HH. PI 3-kinase p110beta: a new target for antithrombotic therapy. Nat Med. 2005 May;11(5):507-14. doi: 10.1038/nm1232. Epub 2005 Apr 17. PMID 15834429